CLINICAL TRIAL: NCT00854035
Title: A Phase III, Randomized, Placebo-Controlled, Double-Blind Clinical Trial and Subsequent Open-Label, Extension Clinical Trial to Study the Efficacy and Safety of Addition of MK-0431/ONO-5435 in Japansese Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Diet/Exercise Therapy and Insulin Monotherapy
Brief Title: MK-0431/ONO-5435 Phase III Clinical Trial - Insulin Add-on Study for Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-5435-15
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: MK-0431/ONO-5435; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- E (Experimental)
  Interventions: Drug: MK-0431/ONO-5435
- P (Placebo Comparator)
  Interventions: Drug: MK-0431/ONO-5435

INTERVENTIONS:
Drug: MK-0431/ONO-5435 — Double-blind period (16 wk); 50 mg QD. The double-blind period will be followed by a 36 wk open-label extension period where MK-0431/ONO-5435 could be titrated from 50mg QD to 100mg QD
  Arms: E
Drug: MK-0431/ONO-5435 — Double-blind period (16 wk); placebo QD. The double-blind period will be followed by a 36 wk open-label extension period where MK-0431/ONO-5435 could be titrated from 50 mg QD to 100 mg QD
  Arms: P

SUMMARY:
This Phase III clinical trial will examine the efficacy, safety, and tolerability of the addition of MK-0431/ONO-5435 to Japanese patients with Type 2 Diabetes Mellitus who have inadequate glycemic control on diet/exercise therapy and insulin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Japanese Patients with Type 2 Diabetes Mellitus who have inadequate glycemic control on diet/exercise therapy and insulin monotherapy

Exclusion Criteria:

* Patients with Type 1 Diabetes Mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
Safety and Tolerability | 16 weeks and 52 weeks

SECONDARY OUTCOMES:
2 hour post-meal glucose | 16 weeks
Fasting plasma glucose | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seki Akiteru, Study Chair — First Division Clinical Development Planning I
Locations (7):
- Japan (7):
  - Chugoku Region, Chugoku
  - Chubu Region, Chūbu
  - Hokuriku Region, Hokuriku
  - Kanto Region, Kanto
  - Kinki Region, Kinki
  - Kyushu Region, Kyushu
  - Tohoku Region, Tōhoku